CLINICAL TRIAL: NCT01816516
Title: Healthy Babies Through Infant Centered Feeding
Acronym: HB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); Colorado State University (Other)
Responsible Party: Principal Investigator, Mildred Horodynski, Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2009-55215-05220
Record Dates: First submitted 2013-03-18; First posted 2013-03-22 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Overweight; Obesity; Infant Overnutrition; Feeding Behavior; Feeding Patterns
Keywords: childhood obesity; low-income; maternal responsiveness; infant feeding; infant feeding practices; infant feeding style; primary prevention
MeSH Terms: conditions — Overweight; Obesity; Infant Nutrition Disorders; Feeding Behavior; Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy Babies (Experimental): Participants receive the Healthy Babies curriculum via 6 in home lessons and 3 follow up telephone calls delivered by Extension paraprofessionals.
  Interventions: Behavioral: Healthy Babies
- EFNEP (Active Comparator): Participants receive the Expanded Food and Nutrition Education Program (EFNEP) curriculum via 6 in home lessons delivered by Extension paraprofessionals.
  Interventions: Behavioral: Expanded Food and Nutrition Education Program

INTERVENTIONS:
Behavioral: Healthy Babies — Each lesson is designed to promote the development of healthy infant eating, and incorporates research-based information, opportunities for mothers to develop and practice skills, and a discussion of strategies to overcome challenges and problem-solving techniques. During lessons, mothers engage in activities in support of lesson goals. Intervention strategies focusing on feeding practices will include modification of the feeding environment (e.g., television off during feeding).
  The telephone contacts, 10 minutes in length, made at 6, 8, and 10 months, reinforce key concepts in the lessons after conclusion of the intervention to maintain effects.
  Arms: Healthy Babies
Behavioral: Expanded Food and Nutrition Education Program — Core EFNEP concepts are United States Department of Agriculture (USDA) My Pyramid, fruits, vegetables, meats, whole grains, food safety, and food resource management. Educators for the EFNEP group will use the EFNEP lessons which address basic knowledge customized for families with infants. Mothers in the EFNEP group will receive a series of six lessons from the nutrition education program offered in each state; they provide a series of lessons focused on nutrition education for families and do not include extensive content on feeding infants.
  Arms: EFNEP

SUMMARY:
Poor feeding practices during infancy contribute to obesity risk because they interfere with infant feeding self-regulation and appropriate growth patterns as infants transition from human milk and/or formula-based diets to solid foods. The goal of the project is to provide an educational intervention that fosters appropriate maternal responsiveness, feeding styles, and feeding practices via infant-centered feeding.

DETAILED DESCRIPTION:
The long-term goal of this integrated project is to contribute to curbing the rising rates of childhood obesity through an effective, multi-component, relationship skill-building and educational intervention that fosters infant-centered feeding to promote appropriate maternal responsiveness, feeding styles, and feeding practices as infants transition to solid foods.

Research Objectives: To evaluate effectiveness of Healthy Babies (HB) compared to the Expanded Food and Nutrition Education Program (EFNEP) at two points in time (when the infant is 6 and 12 months of age) for mothers of infants on maternal responsiveness, feeding style, and feeding practices as infants' transition to solid foods, and to compare infant feeding self-regulation and growth pattern of infants at 6 and 12 months of age between the two groups, HB and EFNEP.

Hypothesis: Compared to mothers of infants who receive traditional EFNEP lessons, mothers who receive HB lessons will achieve an improvement (when the infant is 6 months old that is sustained over time when the infant is 12 months of age) on:

* Maternal responsiveness (measured by appropriately interpreting and responding to infant cues when transitioning their infants to solid foods on the Parent-Child Interaction-Feeding Scale [PCI-F]).
* Maternal feeding styles (measured by feeding beliefs and behaviors on the Infant Feeding Styles Questionnaire).
* Feeding practices (measured by use of appropriate feeding practices when transitioning their infants to solid foods on the PCI-F).

Research Question: How do infants in the HB (intervention) group compare to the infants in the traditional EFNEP group when the infant is 6 and 12 months old on:

* Infant feeding self-regulation (measured by clarity of cues and feeding responsiveness on the PCI-F).
* Infant growth patterns (measured by growth charts).

Extension Objective: To evaluate feasibility, fidelity, and educational effectiveness of the HB intervention. (Process Evaluation)

Research Question: What is the feasibility of integration within Extension by paraprofessionals who deliver HB and for mothers of infants' who receive the HB lessons, related to:

* Paraprofessionals' training, ability to deliver the intervention (fidelity), and satisfaction with the intervention; and
* Mothers' acceptance (recruitment), completion (retention), and satisfaction with the intervention.

Research Question: What is the educational effect of the intervention on maternal knowledge, attitudes, and self-efficacy related to infant feeding?

Research Design. The study will use a randomized clinical trial design in which participants from Michigan (MI) and Colorado (CO) will be randomly assigned to the HB intervention or control (EFNEP) group. The HB intervention, delivered by paraprofessionals (educators), is designed to foster appropriate maternal responsiveness, feeding style, and feeding practices. Participants will be blinded to their group assignment. Data will be collected at three time points by a separate data collection team (not educators): baseline (before the first lesson), follow-up (when infant is six months old), and post follow-up (when infant is 12 months old). These time points have been selected based on the infant's age, such that when an infant is six months old, this is the usual time frame when introducing solid food is recommended to be initiated for all infants, and at 12 months, infants should have an established eating pattern of solid foods. Thus, these points in time were selected rather than immediately following the lessons for consistency in infant age. The age of the infant at time of enrollment will be standardized for timing of the intervention, such that the intervention will begin for all infants between 1 and 4 months of age. Three time points are included to make statistical comparisons and assess the sustainability of changes. Process data will be collected throughout the study.

Participant Recruitment. A total of 546 mother-infant were recruited through community agencies providing services to pregnant women and mothers of infants in Michigan and Colorado (i.e., EFNEP, Breast Feeding Initiative, and Women, Infants and Children's Special Supplemental Nutrition Program for Women, Infants, and Children). Given each state's demographics, Michigan is has a higher proportion of Black minority dyads and Colorado a higher proportion of Hispanic/Latina dyads. Though race/ethnicity/culture is not a specific focus of the study, the sample size will allow us to examine race/ethnic/cultural similarities and differences.

The investigators have recruited of 546 eligible families in MI and CO which will allow for 25% attrition (at each data collection), leaving 278 families at post follow-up (when infant is 12 months old) available for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Mothers aged 18 or older with one, two or three children
* Infants of low-risk births aged birth to 4 months who have not been introduced to solid foods
* Low income (those who qualify for EFNEP, income at or below 185% - 200% of the federal poverty level)
* Infants born between 37 and 42 weeks gestational age with birth weight between 5 pounds 8 ounces and 8 pounds 13 ounces

Exclusion Criteria:

* Male caregivers
* Mothers and/or infants diagnosed with feeding or eating disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 546 (Actual)
Dates: Start 2010-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Maternal Responsiveness at different time points (e.g., 6 months, 12 months) | Change from Baseline in Maternal Responsiveness at 6 months
  Change in maternal responsiveness is measured through an Observational measure (mother-infant feeding interaction): Maternal Responsiveness via Parent-Child Interaction-Feeding Scale (PCI-F) (Formerly Nursing Child Assessment of Feeding Scale)
Change in Baseline in Maternal Responsiveness at different time points (6 months and 12 months) | Change in Baseline in Maternal Responsiveness at 12 months
  Change in Baseline in maternal responsiveness at 12 months is measured via an observational tool: Parent-Child Interaction -Feeding Scale.

SECONDARY OUTCOMES:
Change from Baseline in Feeding Practices assessed at different time points (6 months and 12 months) | Change in Baseline in Feeding Practices at 6 months
  Change in Feeding Practices is assessed via The Infant Feeding Scale (IFS)
Change from Baseline in Feeding Practices assessed at different time points (6 months and 12 months) | Change in Baseline in feeding practices at 12 months
  Change in Baseline in Feeding Practices at 12 months is assessed using the Infant Feeding Scale

OTHER OUTCOMES:
Change from Baseline in Feeding Styles assessed at different times (6 months and 12 months) | Change in Baseline in Feeding Style at 6 months
  Change from Baseline in Feeding Style at 6 months is assessed via the Infant Feeding Styles Questionnaire (IFSQ)
Change from Baseline in Infant Anthropometrics (infant weight and recumbent length) assessed at different time points (6 months and 12 months) | Change in Baseline in infant weight and length in 6 months
  Change from Baseline in Infant weight and recumbent length at 6 months measured using standardized Centers for Disease Control measurement protocol for in-home infant weight and recumbent length.
Change from Baseline in Feeding Style assessed at different time points (6 months and 12 months) | Change in Baseline in Feeding Style at 12 months
  Change from Baseline in Feeding Style at 12 months is assessed using the Infant Feeding Style Questionnaire.
Change from Baseline in infant anthropometrics (infant weight and recumbent length) assessed at different time points (6 months and 12 months) | Change in Baseline in infant weight and recumbent length at 12 months
  Change from Baseline in infant weight and recumbent length at 12 months is assessed using the standardized Centers for Disease Control in-home measurement protocol for infant weight and recumbent length.

CONTACTS AND LOCATIONS:
Overall Officials: Mildred Horodynski, PhD, RN, Principal Investigator — Michigan State University
Locations (2):
- United States (2):
  - Colorado State University, Fort Collins, Colorado
  - Michigan State University, East Lansing, Michigan

REFERENCES:
- [Background] Horodynski MA, Olson B, Baker S, Brophy-Herb H, Auld G, Van Egeren L, Lindau J, Singleterry L. Healthy babies through infant-centered feeding protocol: an intervention targeting early childhood obesity in vulnerable populations. BMC Public Health. 2011 Nov 15;11:868. doi: 10.1186/1471-2458-11-868. PMID 22085421
- [Result] Horodynski MA, Baker S, Van Egeren L, Olson B, Brophy-Herb H, Auld G. The healthy babies curriculum. J Nutr Educ Behav. 2014 Mar-Apr;46(2):151-2. doi: 10.1016/j.jneb.2013.10.002. Epub 2013 Nov 23. No abstract available. PMID 24280320